CLINICAL TRIAL: NCT01073397
Title: Effectiveness of Integral Yoga on Objective and Subjective Menopausal Hot Flashes
Brief Title: Effect of Yoga on Objective and Subjective Menopausal Hot Flashes
Acronym: GLAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00009138; 1R21AT004234-01A2 (NIH)
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Vasomotor Symptoms
Keywords: Menopause; Hot Flashes; Vasomotor symptoms; Yoga
MeSH Terms: conditions — Hot Flashes | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Behavioral (Experimental): Weekly Integral Yoga sessions lasting 90 minutes for 10 weeks with home practice.
  Interventions: Behavioral: Yoga
- Health and Wellness Classes (Active Comparator): Weekly classes on health and wellness lasting 90 minutes for 10 weeks, with additional home practice
  Interventions: Behavioral: Yoga
- Waitlist (No Intervention): This group receives usual care for 10 weeks and is then randomized to one of the study arms.

INTERVENTIONS:
Behavioral: Yoga — Integral Yoga class (90 minutes per class), Once weekly for 10 weeks
  Arms: Behavioral; Health and Wellness Classes

SUMMARY:
The purpose of this research study is to compare yoga and health and wellness classes for helping perimenopausal or newly postmenopausal women who are experiencing hot flashes. The investigators want to learn about the effects of yoga and health and wellness classes on symptoms and other quality of life issues. The results of this study may provide important knowledge to women and clinicians who counsel women with menopausal hot flashes.

DETAILED DESCRIPTION:
Hot flashes and/or night sweats are the most common and troubling symptoms associated with menopause. It is estimated that 64% to 87% of women report experiencing hot flashes for an average of about 4 years. For many women, these symptoms are frequent and severe enough to become debilitating and interfere with daily activities. They often occur at night, disturbing sleep and leading to daytime irritability, fatigue and depressed mood. About 30-40% of menopausal women seek medical help for hot flashes. Relief from hot flashes has been shown to be the primary reason that women initiate hormone therapy (HT).

HT is currently the gold standard for treatment of vasomotor symptoms. A Cochrane Database systematic review showed a 75% reduction in hot flash frequency with hormone therapy compared to placebo.1 However, recent findings from the Women's Health Initiative (WHI) trial indicate that benefits of HT are outweighed by risks, such as coronary heart disease, stroke, pulmonary embolism, breast cancer, and probable dementia. The wide publicity of the WHI results has heightened women's concerns about taking HT and many women have sought alternative treatments for hot flashes. These alternatives include other pharmaceutical agents, herbal or dietary remedies, and behavioral therapies. Unfortunately, many of these agents have a high incidence of side effects or have not been shown to be effective. A recent NIH conference has called for more research on alternative treatments for hot flashes.

Behavioral interventions involving relaxation and slow deep, abdominal breathing have been found to be useful for reducing mild- to moderate-intensity hot flashes. Although the physiological mechanisms for the effectiveness of these interventions are not completely understood, there is some suggestion that they may help reduce sympathetic activity which is related to the narrowing of the thermoneutral zone. It is currently thought that hot flashes are linked to a disruption in thermoregulation and that elevated levels of brain norepinephrine may be the primary mechanism for altered thermoregulation. Breathing techniques form the most integral core of any yoga practice which involves the combination of physical postures (asanas), breathing (pranayama), and deep relaxation (savasana). Despite suggestions that yoga may be beneficial for the relief of hot flashes, these potential benefits have not been well-studied.

To date, treatment efficacy for hot flashes has been limited to self-reported, subjective symptoms. While subjective hot flashes are important from a woman's perspective in her decision-making with respect to treatment, research has shown that they can be influenced by mood and reporting biases. Objective measures are not subject to these biases and have the advantage of providing insight as to whether an intervention has a physiological effect. However, until recently, reliable objective measures that could be used in an ambulatory setting were not available. NCCAM has recently funded the development of new technologies to monitor objective hot flashes in an ambulatory setting, as measured by skin conductance. This technology greatly enhances our ability to fully evaluate the impact of treatment on both subjective and objective hot flashes.

The primary goal of this R21 pilot grant is to obtain preliminary data on the efficacy of Integral Yoga for reducing self-reported menopausal hot flashes. Secondary aims are to determine the impact of yoga on objective hot flashes and other outcomes and study feasibility. Our primary hypothesis will be a greater reduction in subjective hot flash frequency and severity in the yoga group than in two control groups. Secondary outcomes will include a greater reduction in objective hot flash frequency; a greater decrease in hot flash interference; and greater improvement in sleep, other symptoms, mood, perceived stress, and overall quality of life in the yoga group.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 months since last menses
* Age 45-58 years
* Moderate to severe vasomotor symptoms for at least 4 weeks (at least 4/day on average)
* Self-reported general good health
* Adequate English to understand informed consent form, questionnaires, and converse with study staff
* Agree not to use pharmaceutical agents for treating hot flashes during the study

Exclusion Criteria:

* Hormone therapy use within 12 weeks prior to study screening, including systemic estrogen, progestin or androgen therapy
* Selective estrogen receptor modulator (Evista® and Novaldex®) or aromatase inhibitor use within 6 months
* Cancer at any time
* Untreated thyroid disease
* Initiation of herbal or nutritional supplements for hot flashes within the past 4 weeks
* Significant psychiatric disorder, including regular use of antidepressants or anxiolytics
* Regular use of clonidine or Bellergal® within the past 12 weeks
* Any past use of yoga for hot flashes
* Yoga or Acupuncture for any reason within the past 3 months

Ages: 45 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Subjective Hot Flashes | Weekly
  Subjective hot flashes measured by daily diaries

SECONDARY OUTCOMES:
Objective hot flashes | 3 days
  Objective hot flashes measured by skin conductance.
Hot flash interference | 1 week
  This measure assesses the impact of hot flashes on daily activities and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Avis, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States